CLINICAL TRIAL: NCT03768648
Title: Everyday Life Cognition and Non-conventional Magnetic Resonance Markers in RRMS Patients Treated With Aubagio® in a Real-life Setting
Brief Title: Cognition and MRI Markers in MS Patients With Aubagio® Treatment
Acronym: AUBACOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2016/02
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Autoimmune Diseases of the Nervous System; Demyelinating Autoimmune Diseases, CNS; Demyelinating Diseases; Immune System Diseases; Nervous System Diseases; Pathologic Processes; cognitive impairment; ecological assessment; brain MRI
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Autoimmune Diseases of the Nervous System; Demyelinating Autoimmune Diseases, CNS; Demyelinating Diseases; Immune System Diseases; Nervous System Diseases; Pathologic Processes; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient (Experimental): RRMS diagnosis according to McDonald criteria (Polman et al.,2005);
  Interventions: Other: Clinical assessment; Other: Ecological evaluation; Other: Neuropsychological evaluation; Other: Psychological evaluation; Device: MRI Evaluation
- Control (Active Comparator): 40 Healthy controls (HC)
  Interventions: Other: Ecological evaluation; Other: Neuropsychological evaluation; Other: Psychological evaluation; Device: MRI Evaluation

INTERVENTIONS:
Other: Clinical assessment — EDSS (Kurtzke JF; 1983) and the modified MS functional composite (MSFC) score. MS history and MS treatment will be recorded
  Arms: patient
Other: Ecological evaluation — Virtual reality task : Urban DailyCog© and Actual reality
Other: Neuropsychological evaluation — cognitive tests exploring information processing speed, attention/concentration, working and episodic memories and executive function
Other: Psychological evaluation — questionnaires for depression, anxiety and fatigue
Device: MRI Evaluation — morphological MRI and resting state functional MRI (fMRI)

SUMMARY:
Cognitive impairment is nowadays more and more recognized as an important feature of the multiple sclerosis (MS) disease which contributes largely to disability. Cognitive assessment using classical neuropsychological tests are poorly correlated with patient's complaints and daily functioning. Ecological evaluations, recent and innovative way to assess cognitive functions with the true impact of cognitive impairment in everyday daily life of patients. One goal of an ecological test could be to identify MS patients in whom cognitive impairment has a strong interaction with daily life. Different type of ecological evaluation have been recently proposed in MS, including assessment cognitive tasks in a virtual reality environment using the Urban DailyCog® software developed in our laboratory (Hamel et al, 2015). Virtual reality environment assessments are promising in detecting cognitive impairment while providing friendly assessments for patients and simulating daily activities. . Cognitive dysfunction is correlated with white matter diffuse injury in relapsing-remitting MS (RRMS) patients and brain atrophy However, the relationships between structural brain damage and brain connectivity with cognitive functioning assessed by ecological evaluation are also unknown. The use of new techniques for morphological and functional MRI can study the contribution of diffuse white matter (WM) alteration and diffuse gray matter (GM) alterations in cognitive impairment and on their evolution.

The objectives are to evaluate the ecological assessment (Urban DailyCog® and actual reality) to detect cognitive impairment in everyday daily life of patients and their changes and to investigate structural WM and GM damages and the dynamic of functional connectivity for explaining and predicting cognitive disability during two years in RRMS patients treated by the same treatment Aubagio®.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS

* Male or female
* Age 18-60 years
* RRMS diagnosis according to McDonald criteria (Polman et al., 2005);
* Treated with Aubagio® (Indication for first line therapy)
* Native French speaking
* Being affiliated to health insurance
* Having signed an informed consent (at the latest on the day of inclusion and before any examination required by research)

HEALTHY CONTROLS

* Male or Female,
* Age 18-60 years
* Willing to participate and to sign informed consent.
* Being affiliated to health insurance
* Having signed an informed consent (at the latest on the day of inclusion and before any examination required by research)

Exclusion Criteria:

PATIENTS

* History of neurological disease and/or other neurological diseases,
* Psychiatric comorbidity including severe depression according to DSM-IV,
* Alcohol or other addiction to toxic,
* Disabling visual or motor problems preventing participation to neuropsychological assessments,
* Acquisition disorders : Dyslexia, Dysphasia, Dyscalculia and dyspraxia,
* Dosage change, stop or start of hypnotic or anxiolytic or antidepressive treatment less than 30 days
* Relapse since less than one month,
* Steroid treatment less than one month (be taken orally or by infusion) at the dosage of 500mg daily,
* Prior neuropsychological testing with the same tests less than 6 months
* Contra-indication to MRI (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body, claustrophobia) or refusing MRI
* Illiteracy, is unable to count or to read
* Pregnant or breastfeeding women
* Patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent)

HEALTHY CONTROLS

* History of neurological disease and/or neurological diseases
* Psychiatric comorbidity including severe depression according to DSM-IV;
* Alcohol or other toxic addiction;
* Known cognitive complaint or neuropsychological affection
* Hypnotic or anxiolytic or antidepressive treatment,
* Prior neuropsychological testing with the same tests less than 6 months
* Acquisition disorders: Dyslexia, Dysphasia, Dyscalculia and dyspraxia,
* Steroid treatment less than one month (be taken orally or by infusion) at the dosage of 500mg daily,
* Contra-indication to MRI (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body, claustrophobia) or refusing MRI
* Illiteracy, is unable to count or to read
* Pregnant or breastfeeding women
* Person concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Change of composite z ecological score based on individual ecological scores. | At baseline (day 0) and at 24 months from baseline
  The composite z ecological score is the average of z ecological scores of virtual reality task (Urban DailyCog©) and actual reality tests. Z-scores will be calculated for each cognitive score with the following formula: (patient's score - mean value of HC group matched for age, sex, and education level)/standard deviation of the matched HC for each evaluation time (baseline and 2 years).

SECONDARY OUTCOMES:
Change of composite z cognitive score based on individual neuropsychological scores | At baseline (day 0) and at 24 months from baseline
  The composite z cognitive score is the average of z individual cognitive scores. The score from each cognitive test is transformed into z-scores. Z-scores will be calculated for each cognitive score with the following formula: (patient's score - mean value of HC group matched for age, sex, and education level)/standard deviation of the matched HC for each evaluation time. Individual neuropsychological scores included in composite z cognitive score : the Alertness subtest, the divided attention subtest and the visual-scanning subtest from the TAP, The Symbol-digit-modalities-test, the Paced-Auditory-Serial-Addition-Test 3s, reversed span, the Stroop test, the Verbal fluency, Trail Making test, the California Verbal memory learning test and the Brief visual memory test -revised.
Correlation of composite z cognitive score and ecological score with MRI parameters reflecting grey and white matter integrity and anatomic/functional connectivity | At baseline (day 0) and at 24 months from baseline
  The composite z cognitive score and the composite ecological score are the average of z individual cognitive and ecological scores. The score from each cognitive and ecological test is transformed into z-scores. Z-scores will be calculated for each cognitive score with the following formula: (patient's score - mean value of HC group matched for age, sex, and education level)/standard deviation of the matched HC for each evaluation time.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie RUET, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - Service de neurologie, Bordeaux, France